CLINICAL TRIAL: NCT06136533
Title: The Effect of Sarcopenic Obesity on Sleep in Individuals With Obesity Hypoventilation Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Goksen Kuran Aslan, Associated Proffesor, Istanbul University
Other Study IDs: 2023-2/GAslan
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Obesity Hypoventilation Syndrome (OHS); Obesity; Hypoventilation; Respiration Disorders; Sleep Disorder; Breathing-Related; Sarcopenia; Sarcopenic Obesity
Keywords: Obesity Hypoventilation Syndrome (OHS); Obesity; Sarcopenia; Sarcopenic Obesity; Sleep; Quality of Sleep; Sleep Disorder; Breathing-Related; Polysomnography
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Obesity; Hypoventilation; Respiration Disorders; Sleep Wake Disorders; Sarcopenia; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obesity Hypoventilation Syndrome Group: Individuals diagnosed with OHS over the age of 18 years who met the inclusion criteria and who were followed up by Istanbul University Faculty of Medicine, Department of Chest Diseases
  Interventions: Other: Assessment-OHS
- Obesity Hypoventilation Syndrome with Sarcopenic Obesity group: Individuals over the age of 18 years with a diagnosis of OHS and sarcopenic obesity who met the inclusion criteria and who were followed up by Istanbul University Faculty of Medicine, Department of Chest Diseases.
  Interventions: Other: Assessment-Sarcopenic Obesity With OHS

INTERVENTIONS:
Other: Assessment-OHS — Demographic information of individuals diagnosed with OHS without sarcopenia risk is recorded.Bioelectrical Impedance Analysis is used to analyze body composition.The comorbidity levels of the patients were assessed with the 'Modified Charlson Comorbidity Index',sleep quality was assessed with 'Polysomnography' and 'Pittsburgh Sleep Quality Index' and daytime sleepiness was assessed with the 'Epworth Sleepiness Scale'.The assessment of exercise capacity is performed with the 'Six Minute Walking Test' and the assessment of respiratory muscle strength is performed with the 'Electronic Intraoral Pressure Measurement Device'.Patients' physical activity levels are monitored with a pedometer.Quadriceps muscle strength is measured with Hand-held dynamometer and grip strength is measured with Jamar hand dynamometer. The presence of depression is assessed with the 'Beck Depression Inventory' and quality of life with 'Nottingham Health Profile' and 'Functional Outcomes of Sleep Questionnaire'.
  Other Names: Obesity Hypoventilation Syndrome Group
  Groups: Obesity Hypoventilation Syndrome Group
Other: Assessment-Sarcopenic Obesity With OHS — The sarcopenia diagnostic algorithm is used as a reference in the assessment of the presence of sarcopenic obesity. Demographic information of patients diagnosed with sarcopenic obesity is recorded. Then, the comorbidity levels of the patients were assessed with the 'Modified Charlson Comorbidity Index', sleep quality was assessed with 'Polysomnography' and 'Pittsburgh Sleep Quality Index', and daytime sleepiness was assessed with the 'Epworth Sleepiness Scale'. The assessment of exercise capacity is performed with the 'Six Minute Walking Test' and the assessment of respiratory muscle strength is performed with the 'Electronic Intraoral Pressure Measurement Device'. Patients' physical activity levels are monitored with a pedometer. Quadriceps muscle strength is measured with Hand-held dynamometer. The presence of depression is assessed with the 'Beck Depression Inventory' and quality of life with the 'Nottingham Health Profile' and the 'Functional Outcomes of Sleep Questionnaire'.
  Other Names: Obesity Hypoventilation Syndrome with Sarcopenic Obesity group
  Groups: Obesity Hypoventilation Syndrome with Sarcopenic Obesity group

SUMMARY:
Obesity Hypoventilation Syndrome(OHS) is characterized by daytime hypercapnia and sleep-disordered breathing without other causes of hypoventilation in individuals with a body mass index above 30 kg/m2. It is stated that obesity is at the basis of the metabolic changes seen in individuals diagnosed with OHS. Also sedentary lifestyle habits, which are common in obese individuals, cause the risk of sarcopenia due to loss of muscle strength and mass, accumulation of adipose tissue in the body, and decreased exercise capacity. Reduced exercise capacity due to obesity has been shown in the literature to strongly interact with mortality risk. As a result of obesity and all this negative picture, impaired emotional state and decreased quality of life are observed in individuals. Simultaneously, sleep parameters are also negatively affected. In particular, increased adipose tissue leads to loss of muscle mass and strength, increased risk of sarcopenia and sleep-related problems. The association of obesity and sarcopenia is referred to as 'sarcopenic obesity'. Sarcopenic obesity is defined as the coexistence of sarcopenia and obesity. The concept of sarcopenic obesity has recently taken its place in the literature. In particular, there are very few studies on its relationship with sleep parameters. However, while obesity is the basis of OHS, there are no studies on the presence and effects of sarcopenic obesity in this patient group. Based on this point, we aim to investigate the effects of sarcopenic obesity on sleep parameters, exercise capacity and quality of life in individuals with OHS.

DETAILED DESCRIPTION:
Individuals with Obesity Hypoventilation Syndrome followed up in Istanbul University Faculty of Medicine, Department of Chest Diseases will be included in the study. Cases will be divided into two groups according to the presence of sarcopenia. The study will be conducted in accordance with the Declaration of Helsinki and informed consent will be obtained from the patients participating in the study. Before starting the study, the purpose of the study will be explained to the participants and all information about the study will be provided. Patients who agree to participate in the study will be invited to Istanbul University Faculty of Medicine, Department of Chest Diseases on certain days. The sarcopenia diagnostic algorithm is used as a reference in the assessment of the presence of sarcopenic obesity. For the diagnosis of sarcopenic obesity, sarcopenia risk, muscle strength, muscle mass and physical performance level are assessed. Body composition, comorbid levels, sleep and sleep quality, daytime sleepiness, exercise capacity, respiratory muscle strength, peripheral muscle strength, physical activity level, emotional status, sleep-related quality of life and health-related quality of life are assessed in all individuals participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* >50 years old
* 30< BMI< 45 kg/m2
* Patients who have undergone polysomnography evaluation within the last 6 months

Exclusion Criteria:

* Patient who have immobilized for more than 15 days in the last 6 months
* Patient who have used corticosteroids in the last 6 months
* Patient who have been significant weight loss in the last 6 months
* Patient who have been significant serious comorbidities (cognitive impairments, neuromuscular diseases, unstable heart problems, uncontrolled respiratory problems, unresolved thyroid problems, etc.) that may affect participation in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Obesity Hypoventilation Syndrome followed up in Istanbul University Faculty of Medicine, Department of Chest Diseases are included in the study. The subjects are divided into two groups according to the presence of sarcopenia.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Polysomnography (PSG)-Apnea Hypopnea Index | 1 day
  Polysomnography is the gold standard diagnostic method used in the diagnosis of sleep-related respiratory disorders. Polysomnography provides a detailed assessment of sleep. The apnea-hypopnea index (AHI) is the combined average number of apneas and hypopneas that occur per hour of sleep. According to the American Academy of Sleep Medicine (AASM) it is categorized into mild (5-15 events/hour), moderate (15-30 events/hr), and severe (> 30 events/hr). Polysomnography data performed in the last 6 months are recorded to evaluate the apnea hypopnea index of the patients.
Polysomnography (PSG)-Oxygen Desaturation Index | 1 day
  Polysomnography is the gold standard diagnostic method used in the diagnosis of sleep-related respiratory disorders. Polysomnography provides a detailed assessment of sleep. The average number of desaturation episodes per hour is called the oxygen desaturation index (ODI). Desaturation episodes are generally described as a decrease in the mean oxygen saturation of ≥4% (over the last 120 seconds) that lasts for at least 10 seconds. Polysomnography data performed in the last 6 months are recorded to evaluate the oxygen desaturation index of the patients.
Polysomnography (PSG)-Minimum Oxygen Saturation | 1 day
  Polysomnography is the gold standard diagnostic method used in the diagnosis of sleep-related respiratory disorders. Polysomnography provides a detailed assessment of sleep. Polysomnography data performed in the last 6 months are recorded in order to evaluate the minimum oxygen saturation as a percentage.
Polysomnography (PSG)-Oxygen Saturation | 1 day
  Polysomnography is the gold standard diagnostic method used in the diagnosis of sleep-related respiratory disorders. Polysomnography provides a detailed assessment of sleep. Polysomnography data performed in the last 6 months are recorded in order to evaluate the oxygen saturation as a percentage.
Pittsburgh Sleep Quality Index | 1 day
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Developed by researchers at the University of Pittsburgh, the PSQI is intended to be a standardized sleep questionnaire for clinicians and researchers to use with ease and is used for multiple populations. The questionnaire has been used in many settings, including research and clinical activities, and has been used in the diagnosis of sleep disorders.
Nottingham Health Profile | 1 day
  The Nottingham Health Profile (NHP) is a general patient reported outcome measure which seeks to measure subjective health status. It is a questionnaire designed to measure a patient's view of their own health status, in a number of areas. The NHP consists of two parts. The first part focuses on health and comprises 38 items which deal with pain, energy, sleep, mobility, emotional reaction and social isolation. The second part focuses on life areas affected and consists of 7 items which deal with problems regarding occupation, housework, social life, family life, sexual function, hobbies and holidays. The second part of the NHP is optional and can be omitted without ruining the test results.
Functional Outcomes of Sleep Scale (FOSQ) | 1 day
  It is a test used to assess the physical, social and mental impact of excessive daytime sleepiness on activities of daily living. In the Turkish version of the FOSQ, the questions related to sexual activities were excluded and it consists of 26 questions. Each question is evaluated as no difficulty, mild, moderate, moderate, extreme and scored between 0-4 points. A low total score indicates functional insufficiency.
Epworth Sleepiness Scale | 1 day
  Epworth Sleepiness Scale was developed in 1991 by M.W. Developed by Johns. The scale developed to measure sleepiness qualitatively and quantitatively is practical and easy to evaluate and is widely used. Unlike similar scales, it is used to measure the general level of daytime sleepiness. A total score of 11 and above indicates excessive daytime sleepiness. Daytime sleepiness is assessed with this scale.

SECONDARY OUTCOMES:
Modified Charlson Comorbidity Index | 1 day
  The Charlson Comorbidity Index (CCI) was initially developed to predict the survival time of individuals diagnosed with cancer by assigning weights to specific diseases. Today, it is used as a guide for individuals with multiple comorbidities. In this index, diseases are scored based on their morbidity and mortality. The total score is calculated by summing the equivalent scores of diseases. Comorbidity classification is categorized as low (score ≤ 3), moderate (score 4 and 5), high (score 6 and 7), and very high comorbidity (score ≥ 8).
SARC-F Questionnaire | 1 day
  SARC-F is a 5-question questionnaire that asks about strength, assisted walking, getting up from a chair, climbing stairs and falls. Each question is calculated on a "0-2" point scale. A score of zero represents the best score, while a score of ten represents the worst score. Individuals scoring between "0-3" points are considered healthy, while individuals scoring 4 points and above are considered symptomatic. Scores of 4 and above are reported to predict sarcopenia and sarcopenia-related adverse outcomes.
Body Mass Index | 1 day
  Body mass index (BMI) is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Body Fat Percentage | 1 day
  The body fat percentage of a patient is the total mass of fat divided by total body mass, multiplied by 100; body fat includes essential body fat and storage body fat. The body fat percentage of the patients will be evaluated by using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique. And results are recorded in percent.
Body Fluid Percentage | 1 day
  Body fluids, bodily fluids, or biofluids are liquids within the human body. The body fluid percentage of the patients will be evaluated by using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique. And results are recorded in percent.
Muscle Mass | 1 day
  Muscle mass refers to the amount of soft muscle tissue in the body. The muscle mass of the patients will be evaluated by using the "Tanita BC-545N Body Analysis Scale" with the bioelectrical impedance analysis technique. And results are recorded in kg.
Fat-free Muscle | 1 day
  Fat-free mass, sometimes conflated with lean body mass, includes your body's water, organs, bone, and muscle content. In other words, it refers to all of your body components except fat. Fat-free mass is evaluated trough Bioelectrical Impedance Analysis.
Skeletal Muscle Mass | 1 day
  Values changes in total skeletal muscle mass (in kilograms) using bioelectrical impedance analysis and formulas.
Skeletal Muscle Mass Index | 1 day
  Values changes in total skeletal muscle mass index using bioelectrical impedance analysis and formulas.
Anthropometric Measurements-Neck | 1 day
  With the help of a tape measure, neck circumference is measured in cm.
Anthropometric Measurements-Waist | 1 day
  With the help of a tape measure, waist circumference is measured in cm.
Anthropometric Measurements-Abdomen | 1 day
  With the help of a tape measure, abdomen circumference is measured in cm.
Anthropometric Measurements-Hip | 1 day
  With the help of a tape measure, hip circumference is measured in cm.
The Waist-Hip ratio | 1 day
  With the help of a tape measure, waist and hip circumference is measured in cm. Depending on the circumference measurements, waist and hip circumference is calculated as waist to hip ratio.
Six Minutes Walk Test | 1 day
  The distance covered in meters in a straight corridor of 30 meters will be recorded as fast as possible but without running for 6 minutes. The distance that normal individuals should take in this period is 400-700 meters. In addition, oxygen saturation and heart rate, resting fatigue and dyspnea levels will be evaluated with pulse oximetry before and after testing. Modified Borg Dyspnea and Fatigue Scales will be used to determine resting dyspnea and fatigue levels.
The Short Physical Performance Battery (SPPB) | 1 day
  SPPB scale will be used to measure physical function, which is a well-established tool for monitoring function in older people, which contains three kinds of assessments: stand for 10 seconds with feet in 3 different positions, 3-meter or 4-meter walking speed test, and time to rise from a chair for five times. The scores of SPPB range from 0 (worst performance) to 12 (best performance).
Respiratory Muscle Strength | 1 day
  Measurement of respiratory muscle strength will be performed using an electronic mouth pressure measurement device, the "MicroRPM" brand (Micro Medical; UK), in accordance with American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Muscle Strength - Dynamometer | 1 day
  Measurement of respiratory muscle strength will be performed using an electronic mouth pressure measurement device, the "MicroRPM" brand (Micro Medical; UK), in accordance with ATS and ERS criteria.
Physical Activity Level - Pedometer | 1 day
  A pedometer is a small portable device that measures and displays physical activity and counts steps. All patients included in the study use it for 1 week. Each patient will be given 1 pedometer and patients will be asked to record their 1-week data daily on the follow-up chart. It is planned to be used to monitor the daily physical activity level of the patients.
Beck Depression Inventory | 1 day
  Beck Depression Inventory (BDI-II) Scale is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represents a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Goksen KURAN ASLAN, Assoc. Prof., Study Director — Istanbul University - Cerrahpasa; Ece ACIKBAS, PT,MSc, Principal Investigator — Istanbul University - Cerrahpasa; Ozge ERTAN HARPUTLU, PT,MSc, Study Chair — Istanbul University - Cerrahpasa; Melike SARITAS ARSLAN, PT,MSc, Study Chair — Marmara University; Esen KIYAN, Prof., Study Chair — Istanbul University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No